CLINICAL TRIAL: NCT01540045
Title: Effect of Chemotherapy With Paclitaxel and Cisplatin on Development Dysgeusia in Non-small Cell Lung Cancer Patients
Brief Title: Effect of Chemotherapy With Paclitaxel/Cisplatin on Development Dysgeusia in Non Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez, Head Of the Thoracic Oncology Clinic. SNI II, Instituto Nacional de Cancerologia de Mexico
Other Study IDs: ECPCDLC2012
Record Dates: First submitted 2012-01-13; First posted 2012-02-28 (Estimated); Results first posted 2015-03-18 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Non-Small Cell Lung Cancer; Dysgeusia; Taste Disorders; Lung Neoplasms; Small Cell Lung Carcinoma
Keywords: Non-Small Cell Lung Cancer; Dysgeusia; Antineoplastic Combined Chemotherapy Protocols; Paclitaxel; Cisplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Dysgeusia; Taste Disorders; Lung Neoplasms; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- BASELINE: Outpatients from National Cancer Institute with stage III and IV NSCLC candidates for 1 st line chemotherapy paclitaxel-cisplatin based agreeing to participate in the study

SUMMARY:
One of the most widely used treatments for non-small cell lung cancer (NSCLC) is the combination of paclitaxel-cisplatin. These drugs may contribute to taste alterations like dysgeusia. Which alters the feeding of cancer patients, contributing to the anorexia, weight loss and malnutrition, which leads to a prognostic impact in a lower patient response to chemotherapy, radiotherapy and surgical treatment as well as increased toxic effects, impacting treatment discontinuation and therefore, morbidity and survival of patients. The objective of this study is to describe the threshold of perception and recognition of basic tastes in patients with NSCLC before treatment with platin and paclitaxel-based chemotherapy and after the second cycle, and analyze the effect in the developement of dysgeusia, as well as the association between these and the nutritional status and quality of life.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of death from malignancies in our country. It was recently reported to induce 11.5% of cancer deaths in Mexico, with a rate of 6.5 per 100 000 people.

Non-Small Cell Lung Cancer (NSCLC) accounts for 80% of all lung cancer cases. Less than 20% has resectable disease and in the National Cancer Institute of Mexico exclusively less than 2%, representing chemotherapy the standard of care in these patients.

One of the most widely used drug combinations is paclitaxel-cisplatin. It has been reported a prevalence of malnutrition in 60 to 79% in this type of cancer, being the major contributor to morbidity and mortality. The etiology resides both in the systemic effects of the tumor and toxic effects of treatment as low levels hematologic, nausea, vomiting, mucositis, anorexia, dysgeusia, among others.

Weight loss has a strong impact on the response to chemotherapy, radiotherapy and surgery, as well as increased toxic effects impacting the discontinuation of treatment and is considered an independent predictor of survival for most patients with NSCLC. Is estimated that over 20% of cancer patients the cause of death are inanition effects.

Among the most frequent symptoms in advanced unresectable cancer or its treatment that may affect food intake and hence nutritional status, are the early satiety and dysgeusia (61% and 46% respectively). As are difficult to change early satiety, dysgeusia is a field for selecting strategies in its management.

The dysgeusia is defined as a change in taste that can manifest as a distortion of taste, lack of taste (ageusia), decreased sensitivity of perception (hypogeusia) or increased sensitivity to some or all flavors (hypergeusia).

The development of dysgeusia have clinical significance in the etiology of cancer anorexia because it can affect eating habits and contribute to weight loss or malnutrition and consequently affect the quality of life.

The chemotherapy may contribute to dysgeusia. It has reported a prevalence of 56.3% of Dysgeusia in cancer patients under this type of treatment. As well, zinc deficiency has been associated with the hypogeusia, this metal to be involved at various levels in the physiology of the role of taste at various levels of cell several organization.

Several studies have linked consumption dysgeusia with energy and macronutrients, weight loss, lack of appetite and early satiety.

The type of tumor, stage, chemotherapy regimen and serum zinc levels are associated with dysgeusia, but the exact mechanism underlining these disturbances are not known at totality. No known if chemotherapy or before this is presented dysgeusia. In addition there are few studies in this area and with methodological weaknesses, among which include heterogeneous population (patients with a diagnosis of malignancy of breast, lung, prostate, multiple myeloma and lymphoma), different patterns of treatment(different chemotherapy drugs, radiotherapy schedules and combination of both forms of measurement of dysgeusia, besides the absence of dysgeusia baseline evaluation before chemotherapy to establish a causal association between chemotherapy and taste alteration.

Also, is unknown if dysgeusia impact on body composition determined by bioelectrical impedance, phase angle in and consumption of micronutrients (iron, sodium, zinc, B6, B12).

That's why is necessary to continue studying this phenomenon to develop a better understanding of the nature, frequency, severity and duration of dysgeusia in patients with advanced lung cancer, the role that zinc exerts in its development and its impact on consumption food, anthropometric parameters and quality of life in such patients before and after chemotherapy in the same regimen of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old with INCan histopathological diagnosis of Lung Cancer Stage III or IV
* ECOG score ≤ 2
* Candidates for first-line chemotherapy based 1 st Paclitaxel / cisplatin 200 mg/m2 and 75 every 3 weeks
* Signed informed consent (and ethical scientific committee No. (010/023 (IMO) (CB/618

Exclusion Criteria:

* Patients who withdraw their consent and not want to continue with the evaluation of the study
* Common cold or hay fever, recent dental procedure, evidence of gingival inflammation or infection or oral mucosa
* People diagnosed with epilepsy or some other neurological disorders associated
* Concomitant radiotherapy in head and neck.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients from National Cancer Institute with stage III and IV NSCLC candidates for 1 st line chemotherapy paclitaxel-cisplatin based agreeing to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar G Arrieta, MD M Sc, Principal Investigator — Mexico. Nacional Cancer Institute
Locations (1):
- National Cancer Institute of Mexico, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Ruiz-Godoy L, Rizo Rios P, Sanchez Cervantes F, Osornio-Vargas A, Garcia-Cuellar C, Meneses Garcia A. Mortality due to lung cancer in Mexico. Lung Cancer. 2007 Nov;58(2):184-90. doi: 10.1016/j.lungcan.2007.06.007. Epub 2007 Jul 30. PMID 17659812
- [Background] Sarhill N, Mahmoud FA, Christie R, Tahir A. Assessment of nutritional status and fluid deficits in advanced cancer. Am J Hosp Palliat Care. 2003 Nov-Dec;20(6):465-73. doi: 10.1177/104990910302000610. PMID 14649565
- [Background] Wie GA, Cho YA, Kim SY, Kim SM, Bae JM, Joung H. Prevalence and risk factors of malnutrition among cancer patients according to tumor location and stage in the National Cancer Center in Korea. Nutrition. 2010 Mar;26(3):263-8. doi: 10.1016/j.nut.2009.04.013. Epub 2009 Aug 8. PMID 19665873
- [Background] Arrieta O, Michel Ortega RM, Villanueva-Rodriguez G, Serna-Thome MG, Flores-Estrada D, Diaz-Romero C, Rodriguez CM, Martinez L, Sanchez-Lara K. Association of nutritional status and serum albumin levels with development of toxicity in patients with advanced non-small cell lung cancer treated with paclitaxel-cisplatin chemotherapy: a prospective study. BMC Cancer. 2010 Feb 21;10:50. doi: 10.1186/1471-2407-10-50. PMID 20170547
- [Background] Halyard MY. Taste and smell alterations in cancer patients--real problems with few solutions. J Support Oncol. 2009 Mar-Apr;7(2):68-9. No abstract available. PMID 19408460
- [Background] Hong JH, Omur-Ozbek P, Stanek BT, Dietrich AM, Duncan SE, Lee YW, Lesser G. Taste and odor abnormalities in cancer patients. J Support Oncol. 2009 Mar-Apr;7(2):58-65. PMID 19408458
- [Background] Rolls ET. The representation of umami taste in the taste cortex. J Nutr. 2000 Apr;130(4S Suppl):960S-5S. doi: 10.1093/jn/130.4.960S. PMID 10736361
- [Background] Comeau TB, Epstein JB, Migas C. Taste and smell dysfunction in patients receiving chemotherapy: a review of current knowledge. Support Care Cancer. 2001 Nov;9(8):575-80. doi: 10.1007/s005200100279. PMID 11762967
- [Background] Arrieta O, Hernandez-Pedro N, Fernandez-Gonzalez-Aragon MC, Saavedra-Perez D, Campos-Parra AD, Rios-Trejo MA, Ceron-Lizarraga T, Martinez-Barrera L, Pineda B, Ordonez G, Ortiz-Plata A, Granados-Soto V, Sotelo J. Retinoic acid reduces chemotherapy-induced neuropathy in an animal model and patients with lung cancer. Neurology. 2011 Sep 6;77(10):987-95. doi: 10.1212/WNL.0b013e31822e045c. Epub 2011 Aug 24. PMID 21865574
- [Background] Bernhardson BM, Tishelman C, Rutqvist LE. Self-reported taste and smell changes during cancer chemotherapy. Support Care Cancer. 2008 Mar;16(3):275-83. doi: 10.1007/s00520-007-0319-7. Epub 2007 Aug 21. PMID 17710445
- [Background] Gupta D, Lammersfeld CA, Vashi PG, King J, Dahlk SL, Grutsch JF, Lis CG. Bioelectrical impedance phase angle in clinical practice: implications for prognosis in stage IIIB and IV non-small cell lung cancer. BMC Cancer. 2009 Jan 28;9:37. doi: 10.1186/1471-2407-9-37. PMID 19175932
- [Background] Hernandez-Avila M, Romieu I, Parra S, Hernandez-Avila J, Madrigal H, Willett W. Validity and reproducibility of a food frequency questionnaire to assess dietary intake of women living in Mexico City. Salud Publica Mex. 1998 Mar-Apr;40(2):133-40. doi: 10.1590/s0036-36341998000200005. PMID 9617194
- [Background] Thoresen L, Fjeldstad I, Krogstad K, Kaasa S, Falkmer UG. Nutritional status of patients with advanced cancer: the value of using the subjective global assessment of nutritional status as a screening tool. Palliat Med. 2002 Jan;16(1):33-42. doi: 10.1191/0269216302pm486oa. PMID 11963449
- [Background] Bauer J, Capra S, Ferguson M. Use of the scored Patient-Generated Subjective Global Assessment (PG-SGA) as a nutrition assessment tool in patients with cancer. Eur J Clin Nutr. 2002 Aug;56(8):779-85. doi: 10.1038/sj.ejcn.1601412. PMID 12122555
- [Background] Muscaritoli M, Anker SD, Argiles J, Aversa Z, Bauer JM, Biolo G, Boirie Y, Bosaeus I, Cederholm T, Costelli P, Fearon KC, Laviano A, Maggio M, Rossi Fanelli F, Schneider SM, Schols A, Sieber CC. Consensus definition of sarcopenia, cachexia and pre-cachexia: joint document elaborated by Special Interest Groups (SIG) "cachexia-anorexia in chronic wasting diseases" and "nutrition in geriatrics". Clin Nutr. 2010 Apr;29(2):154-9. doi: 10.1016/j.clnu.2009.12.004. Epub 2010 Jan 8. PMID 20060626
- [Background] Halyard MY, Jatoi A, Sloan JA, Bearden JD 3rd, Vora SA, Atherton PJ, Perez EA, Soori G, Zalduendo AC, Zhu A, Stella PJ, Loprinzi CL. Does zinc sulfate prevent therapy-induced taste alterations in head and neck cancer patients? Results of phase III double-blind, placebo-controlled trial from the North Central Cancer Treatment Group (N01C4). Int J Radiat Oncol Biol Phys. 2007 Apr 1;67(5):1318-22. doi: 10.1016/j.ijrobp.2006.10.046. PMID 17394940
- [Result] Brennan MT, Elting LS, Spijkervet FK. Systematic reviews of oral complications from cancer therapies, Oral Care Study Group, MASCC/ISOO: methodology and quality of the literature. Support Care Cancer. 2010 Aug;18(8):979-84. doi: 10.1007/s00520-010-0856-3. Epub 2010 Mar 20. PMID 20306090
- [Result] Gallagher P, Tweedle DE. Taste threshold and acceptability of commercial diets in cancer patients. JPEN J Parenter Enteral Nutr. 1983 Jul-Aug;7(4):361-3. doi: 10.1177/0148607183007004361. PMID 6413712
- [Result] Mattes RD, Cowart BJ, Schiavo MA, Arnold C, Garrison B, Kare MR, Lowry LD. Dietary evaluation of patients with smell and/or taste disorders. Am J Clin Nutr. 1990 Feb;51(2):233-40. doi: 10.1093/ajcn/51.2.233. PMID 2305710
- [Result] Hutton JL, Baracos VE, Wismer WV. Chemosensory dysfunction is a primary factor in the evolution of declining nutritional status and quality of life in patients with advanced cancer. J Pain Symptom Manage. 2007 Feb;33(2):156-65. doi: 10.1016/j.jpainsymman.2006.07.017. PMID 17280921
- [Result] Rehwaldt M, Wickham R, Purl S, Tariman J, Blendowski C, Shott S, Lappe M. Self-care strategies to cope with taste changes after chemotherapy. Oncol Nurs Forum. 2009 Mar;36(2):E47-56. doi: 10.1188/09.onf.e47-e56. PMID 19273394
- [Result] Steinbach S, Hummel T, Bohner C, Berktold S, Hundt W, Kriner M, Heinrich P, Sommer H, Hanusch C, Prechtl A, Schmidt B, Bauerfeind I, Seck K, Jacobs VR, Schmalfeldt B, Harbeck N. Qualitative and quantitative assessment of taste and smell changes in patients undergoing chemotherapy for breast cancer or gynecologic malignancies. J Clin Oncol. 2009 Apr 10;27(11):1899-905. doi: 10.1200/JCO.2008.19.2690. Epub 2009 Mar 16. PMID 19289621
- [Result] Zabernigg A, Gamper EM, Giesinger JM, Rumpold G, Kemmler G, Gattringer K, Sperner-Unterweger B, Holzner B. Taste alterations in cancer patients receiving chemotherapy: a neglected side effect? Oncologist. 2010;15(8):913-20. doi: 10.1634/theoncologist.2009-0333. Epub 2010 Jul 28. PMID 20667968
- [Result] Sanchez-Lara K, Sosa-Sanchez R, Green-Renner D, Rodriguez C, Laviano A, Motola-Kuba D, Arrieta O. Influence of taste disorders on dietary behaviors in cancer patients under chemotherapy. Nutr J. 2010 Mar 24;9:15. doi: 10.1186/1475-2891-9-15. PMID 20334666
- [Result] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Derived] Turcott JG, Juarez-Hernandez E, De la Torre-Vallejo M, Sanchez-Lara K, Luvian-Morales J, Arrieta O. Value: Changes in the Detection and Recognition Thresholds of Three Basic Tastes in Lung Cancer Patients Receiving Cisplatin and Paclitaxel and Its Association with Nutritional and Quality of Life Parameters. Nutr Cancer. 2016;68(2):241-9. doi: 10.1080/01635581.2016.1144075. Epub 2016 Mar 4. PMID 26943275

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruit patients since September 2010 to July 2012
Pre-assignment Details: We invited to participate 40 patients who completed their baseline evaluation and their follow up after two cycles of chemotherapy using paclitaxel (175 mg/m2) and cisplatin (75 mg/m2). The main reason of exclusion was death followed by not returning to the institution.
Groups:
- Pre-chemotherapy Patientes =40: Outpatients from National Cancer Institute with stage III and IV NSCLC candidates for 1 st line chemotherapy paclitaxel-cisplatin based agreeing to participate in the study
Period: Overall Study
Arm/Group | Pre-chemotherapy Patientes =40
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: We invited to participate 72 patients with NSCLC newly diagnosed, but only 40 patients completed their baseline evaluation and their follow up after two cycles of chemotherapy using paclitaxel (175 mg/m2) and cisplatin (75 mg/m2). The main reason of exclusion was death followed by not returning to the institution.
Arm/Group | Pre-chemotherapy Patientes =40
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20
Region of Enrollment [Number; unit: participants]
  Mexico | 40

OUTCOME MEASURES:

1. Primary Outcome: Dysgeusia (UMAMI Perception)
Description: Describe the threshold of perception and recognition (PT and RT, respectively) umami) with 5 dilutions with different concentrations.
  The patients were instructed to taste each 5 ml dilution in ascending order and to rinse the dilution around the entire oral cavity. After each rinse, the patients were asked whether the sample they took tasted different from water to identify their PT, which was assigned to the lowest concentration at which the subject perceived a difference in taste from water. If so, then the patients were asked to identify the taste to define their RT, which was assigned to the lowest concentration at which the subject identified the taste.
Time Frame: Change from Baseline in threshold of perception at 6 weeks
Measure: Median (Full Range); unit: μmol/ml
Groups:
- Pre-chemotherapy Patientes: measurement pre-chemotherapy
- Post-chemotherapy Patients: measurement post-chemotherapy
Arm/Group | Pre-chemotherapy Patientes | Post-chemotherapy Patients
Number analyzed (Participants) | 40 | 39
μmol/ml | .3 [.3 to 3.3] | .3 [.3 to 2.7]
Statistical Analysis 1: Comparison: Pre-chemotherapy Patientes vs Post-chemotherapy Patients; For the paired analysis of taste acuity we used Wilcoxon for difference between baseline and 6 weeks later; Test type: Superiority or Other; p = 0.013, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: BODY COMPOSITION
Description: fat mass and lean body mass pre-post chemotherapy
Time Frame: Change from Baseline in perception and recognition thresholds at 6 weeks
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Pre-chemotherapy Patientes: body composition pre-chemotherapy
- Post-chemotherapy Patients: body composition post chemotherapy
Arm/Group | Pre-chemotherapy Patientes | Post-chemotherapy Patients
Number analyzed (Participants) | 40 | 40
kg
  FAT MASS (kg) | 20.09 (7.7) | 19.67 (6.5)
  LEAN BODY MASS (kg) | 41.79 (13) | 41.26 (11.9)
Statistical Analysis 1: Comparison: Pre-chemotherapy Patientes vs Post-chemotherapy Patients; we evaluated body fat before and after 2 cycles of cisplatin/paclitaxel based chemotheprapy; Test type: Superiority or Other; p = 0.671, t-test, 2 sided
Statistical Analysis 2: Comparison: Pre-chemotherapy Patientes vs Post-chemotherapy Patients; we evaluated lean body mass before and after 2 cycles of cisplatin/paclitaxel based chemotheprapy; Test type: Superiority or Other; p = 0.694, t-test, 2 sided

3. Secondary Outcome: Body Mass Index
Description: Body mass index, using the formula kg/m^2
Time Frame: Change from Baseline in threshold of perception and recognition at 6 weeks
Measure: Mean (Standard Deviation); unit: kg/m^2
Groups:
- Pre-chemotherapy Patientes: body mass index pre-chemotherapty
- Post-chemotherapy Patients: body mass index post chemotherapy
Arm/Group | Pre-chemotherapy Patientes | Post-chemotherapy Patients
Number analyzed (Participants) | 40 | 40
kg/m^2 | 24.5 (4) | 24.1 (4)
Statistical Analysis 1: Comparison: Pre-chemotherapy Patientes vs Post-chemotherapy Patients; Test type: Superiority or Other; p = 0.118, t-test, 2 sided

4. Secondary Outcome: Subjective Global Assessment
Description: validated questionnaire to identify patients with malnutrition or risk of malnutrition Subjective global assessment (PG-SGA) was used to assess and classify patients as having severe or moderate malnourishment (B or C) or as being well nourished (A).
Time Frame: descriptive values before chemotherapy
Measure: Number; unit: participants
Groups:
- Pre-chemotherapy Patientes: Subjective Global Assessment pre-chemotherapy
- Post-chemotherapy Patientes: Subjective Global Assessment post chemotherapy
Arm/Group | Pre-chemotherapy Patientes | Post-chemotherapy Patientes
Number analyzed (Participants) | 40 | 40
participants
  SGA A | 26 | 23
  SGA B & C | 14 | 17
Statistical Analysis 1: Comparison: Pre-chemotherapy Patientes vs Post-chemotherapy Patientes; Subjective global assessment (PG-SGA) was used to assess and classify patients as having severe or moderate malnourishment (B or C) or as being well nourished (A); Test type: Superiority or Other; p = 0.607, McNemar

5. Secondary Outcome: PROTEIN AND FAT Consumption
Description: energy and nutrimental consumption was estimated by questionnaire SNUT difference between ≥ Sweet perception thresholds vs < Sweet perception thresholds after chemotherapy
Time Frame: participants were evaluated baseline and after 2 cycles of chemotherapy, an average of 6 weeks
Measure: Mean (Standard Deviation); unit: gr
Groups:
- ≥ Sweet Perception Thresholds After Chemotherapy: patient with more sensibility to perceive sweet taste from food
- < Sweet Perception Thresholds After Chemotherapy: patient with less sensibility to perceive sweet taste from food
Arm/Group | ≥ Sweet Perception Thresholds After Chemotherapy | < Sweet Perception Thresholds After Chemotherapy
Number analyzed (Participants) | 29 | 11
gr
  proteins | 59.12 (32.7) | 91.07 (33.1)
  animal proteins | 28.2 (14) | 49.29 (18.5)
  fat | 60.1 (26.2) | 91.77 (31.6)
Statistical Analysis 1: Comparison: ≥ Sweet Perception Thresholds After Chemotherapy vs < Sweet Perception Thresholds After Chemotherapy; protein consumption was estimated by questionnaire SNUT difference between ≥ Sweet perception thresholds compared to < Sweet perception thresholds after chemotherapy; Test type: Superiority or Other; p = 0.015, t-test, 2 sided
Statistical Analysis 2: Comparison: ≥ Sweet Perception Thresholds After Chemotherapy vs < Sweet Perception Thresholds After Chemotherapy; animal protein consumption was estimated by questionnaire SNUT difference between ≥ Sweet perception thresholds vs < Sweet perception thresholds after chemotherapy; Test type: Superiority or Other; p = 0.010, t-test, 2 sided
Statistical Analysis 3: Comparison: ≥ Sweet Perception Thresholds After Chemotherapy vs < Sweet Perception Thresholds After Chemotherapy; FAT consumption was estimated by questionnaire SNUT difference between ≥ Sweet perception thresholds vs < Sweet perception thresholds after chemotherapy; Test type: Superiority or Other; p = 0.004, t-test, 2 sided

6. Secondary Outcome: IRON Consumption
Description: IRON consumption was estimated by questionnaire SNUT difference between ≥ Sweet perception thresholds vs < Sweet perception thresholds after chemotherapy
Time Frame: participants were evaluated baseline and after 2 cycles of chemotherapy, an average of 6 weeks
Measure: Mean (Standard Deviation); unit: mg
Groups:
- ≥ Sweet Perception Thresholds After Chemotherapy: IRON CONSUMPTION ≥ Sweet perception thresholds after chemotherapy
- < Sweet Perception Thresholds After Chemotherapy: IRON CONSUMPTION < Sweet perception thresholds after chemotherapy
Arm/Group | ≥ Sweet Perception Thresholds After Chemotherapy | < Sweet Perception Thresholds After Chemotherapy
Number analyzed (Participants) | 29 | 11
mg | 10.8 (7.5) | 16.11 (6.3)

7. Primary Outcome: Dysgeusia (UMAMI Recognition)
Description: Describe the threshold recognition (RT) of umami with 5 dilutions with different concentrations.
  The patients were instructed to taste each 5 ml dilution in ascending order and to rinse the dilution around the entire oral cavity. After each rinse, the patients were asked whether the sample they took tasted different from water to identify their PT, which was assigned to the lowest concentration at which the subject perceived a difference in taste from water. If so, then the patients were asked to identify the taste to define their RT, which was assigned to the lowest concentration at which the subject identified the taste.
Time Frame: Change from Baseline in threshold of perception at 6 weeks
Population: For the paired analysis of taste acuity we used Wilcoxon for difference between baseline and 6 weeks later.
Measure: Median (Full Range); unit: μmol/ml
Arm/Group | Pre-chemotherapy Patientes | Post-chemotherapy Patients
Number analyzed (Participants) | 40 | 39
μmol/ml | 2.4 [.3 to 3.3] | 1.5 [.3 to 3.3]
Statistical Analysis 1: Comparison: Pre-chemotherapy Patientes vs Post-chemotherapy Patients; For the paired analysis of taste acuity we used Wilcoxon for difference between baseline and 6 weeks later; Test type: Superiority or Other; p = 0.28, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Quality o f Life
Description: The HRQL evaluation was assessed using the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaires specific for cancer and for LC (EORTC-QLQ-C30 and QLQ-LC13). [18, 19] Scores for the multi-item functional or symptom scales and the single items scales were calculated using a linear transformation of raw scores to produce a range from 0 to 100, as described by EORTC. A score of 100 represents the best score for the global health status and functional scales of QoL or 0 in the symptom rating.
Time Frame: participants were evaluated baseline and after 2 cycles of chemotherapy, an average of 6 weeks
Measure: Median (Full Range); unit: Scores on a scale
Groups:
- HRQL Pre-chemotherapy; HRQL Post-chemotherapy: Score of scale HRQL EORTC
Arm/Group | HRQL Pre-chemotherapy | HRQL Post-chemotherapy
Number analyzed (Participants) | 40 | 40
Scores on a scale
  Global status | 58.33 [0 to 100] | 66.67 [0 to 100]
  Role functioning | 66.67 [0 to 100] | 83.33 [0 to 100]
  Emotional functioning | 66.67 [0 to 100] | 91.67 [0 to 100]
  Fatigue | 38.8 [0 to 100] | 22.22 [0 to 100]
  Appetite loss | 33.33 [0 to 100] | 0 [0 to 100]
  Constipation | 33.33 [0 to 100] | 0 [0 to 100]
Statistical Analysis 1: Comparison: HRQL Pre-chemotherapy vs HRQL Post-chemotherapy; change in status global of quality of life between ≤ compared to > umami recognition threshold after chemotherapy by EORT questionnaire; Test type: Superiority or Other; p = 0.889, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: HRQL Pre-chemotherapy vs HRQL Post-chemotherapy; change in functional role of quality of life between ≤ compared to > umami recognition threshold after chemotherapy by EORT questionnaire; Test type: Superiority or Other; p = 0.293, Wilcoxon (Mann-Whitney) — clinically significant
Statistical Analysis 3: Comparison: HRQL Pre-chemotherapy vs HRQL Post-chemotherapy; change in emotional functioning of quality of life between ≤ compared to > umami recognition threshold after chemotherapy by EORT questionnaire; Test type: Superiority or Other; p = 0.009, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: HRQL Pre-chemotherapy vs HRQL Post-chemotherapy; change in fatigue scale of quality of life between ≤ compared to > umami recognition threshold after chemotherapy by EORT questionnaire; Test type: Superiority or Other; p = 0.213, Wilcoxon (Mann-Whitney) — clinically significant
Statistical Analysis 5: Comparison: HRQL Pre-chemotherapy vs HRQL Post-chemotherapy; change in appetite loss of quality of life between ≤ compared to > umami recognition threshold after chemotherapy by EORT questionnaire; Test type: Superiority or Other; p = 0.595, Wilcoxon (Mann-Whitney) — clinically significant
Statistical Analysis 6: Comparison: HRQL Pre-chemotherapy vs HRQL Post-chemotherapy; change in constipation scale of quality of life between ≤ compared to > umami recognition threshold after chemotherapy by EORT questionnaire; Test type: Superiority or Other; p = 0.068, Wilcoxon (Mann-Whitney) — clinically significant

9. Secondary Outcome: Change From Baseline in Albumin After 2 Cycles of Chemotherapy
Description: comparison of patients who increased or decreased their sensibility to the PT of umami taste
Time Frame: participants were evaluated baseline and after 2 cycles of chemotherapy, an average of 6 weeks
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- > or = Umami Perception Thresholds: patients with more or the same sensibility to umami taste pre-post chemotherapy in NSCLC patients.
  (> UPT) = more sensibility to umami perception
- < Umami Perception Thresholds: patients with less sensibility to umami taste pre-post chemotherapy in NSCLC patients.
  (< UPT) = less sensibility to umami perception
Arm/Group | > or = Umami Perception Thresholds | < Umami Perception Thresholds
Number analyzed (Participants) | 34 | 6
g/dL | -0.4 (0.11) | 0.28 (0.1)
Statistical Analysis 1: Comparison: > or = Umami Perception Thresholds vs < Umami Perception Thresholds; Test type: Superiority or Other; p = 0.05, t-test, 2 sided

10. Secondary Outcome: Peripheral Neuropathy (QLQ-C30 Version 3, EORTC)
Description: comparison of peripheral neuropathy patients who increased or decreased their sensibility to the PT of umami taste The HRQL evaluation was assessed using the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaires specific for cancer and for LC (EORTC-QLQ-C30 and QLQ-LC13). Scores for the multi-item functional or symptom scales and the single items scales were calculated using a linear transformation of raw scores to produce a range from 0 to 100, as described by EORTC. A score of 100 represents the best score for the global health status and functional scales of QoL or 0 in the symptom rating.
Time Frame: participants were followed for the duration of 2 cycles of chemotherapy, an average of 6 weeks
Measure: Median (Full Range); unit: Units on a scale
Groups:
- > or = Umami Perception Thresholds: peripheral neuropathy in patients with more or the same sensibility to umami taste pre-post chemotherapy in NSCLC patients.
  (> UPT) = more sensibility to umami perception
- < Umami Perception Thresholds: peripheral neuropathy patients with less sensibility to umami taste pre-post chemotherapy in NSCLC patients.
  (< UPT) = less sensibility to umami perception
Arm/Group | > or = Umami Perception Thresholds | < Umami Perception Thresholds
Number analyzed (Participants) | 30 | 6
Units on a scale | 33.33 [0 to 100] | 16.66 [0 to 66.67]
Statistical Analysis 1: Comparison: > or = Umami Perception Thresholds vs < Umami Perception Thresholds; change in peripheral neuropathy scale of quality of life between > ó = compared to < umami recognition threshold after chemotherapy by EORT questionnaire; Test type: Superiority or Other; p = 0.240, Wilcoxon (Mann-Whitney) — clinically significant

11. Secondary Outcome: Global Status of Quality of Life (C-30,LC13 EORTC)
Description: differences in global status of QoL scale (C-30,LC13 EORTC) between those with more or less sensibility to recognize the umami taste.
  score of scale 0-100, a higher score represents better overall state.
Time Frame: time between baseline and before 2 cycles of chemotherapy, an average of 6 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- < or = Umami Recognition Thresholds; > Umami Recognition Thresholds: quality of life scales in patient with more or the same sensibility to recognize the umami taste
Arm/Group | < or = Umami Recognition Thresholds | > Umami Recognition Thresholds
Number analyzed (Participants) | 20 | 9
units on a scale | 75 [1.66 to 99.58] | 66.67 [8.33 to 100]
Statistical Analysis 1: Comparison: < or = Umami Recognition Thresholds vs > Umami Recognition Thresholds; change in status global of quality of life between > ó = compared to < umami recognition threshold after chemotherapy by EORT questionnaire; Test type: Superiority or Other; p = 0.036, Wilcoxon (Mann-Whitney)

12. Primary Outcome: Dysgeusia (SWEET Perception)
Description: Describe the threshold perception (PT) of sweet taste with 5 dilutions with different concentrations.
  The patients were instructed to taste each 5 ml dilution in ascending order and to rinse the dilution around the entire oral cavity. After each rinse, the patients were asked whether the sample they took tasted different from water to identify their PT, which was assigned to the lowest concentration at which the subject perceived a difference in taste from water. If so, then the patients were asked to identify the taste to define their RT, which was assigned to the lowest concentration at which the subject identified the taste.
Time Frame: Change from Baseline in threshold of perception at 6 weeks
Population: For the paired analysis of taste acuity we used Wilcoxon for difference between baseline and 6 weeks later.
Measure: Median (Full Range); unit: μmol/ml
Arm/Group | Pre-chemotherapy Patientes | Post-chemotherapy Patients
Number analyzed (Participants) | 40 | 39
μmol/ml | 3.5 [3.5 to 18.5] | 3.5 [3.5 to 18.5]
Statistical Analysis 1: Comparison: Pre-chemotherapy Patientes vs Post-chemotherapy Patients; For the paired analysis of taste acuity we used Wilcoxon for difference between baseline and 6 weeks later; Test type: Superiority or Other; p = 0.312, Wilcoxon (Mann-Whitney)

13. Primary Outcome: Dysgeusia (SWEET Recognition)
Description: Describe the recognition threshold (RT) of sweet taste with 5 dilutions with different concentrations.
  The patients were instructed to taste each 5 ml dilution in ascending order and to rinse the dilution around the entire oral cavity. After each rinse, the patients were asked whether the sample they took tasted different from water to identify their PT, which was assigned to the lowest concentration at which the subject perceived a difference in taste from water. If so, then the patients were asked to identify the taste to define their RT, which was assigned to the lowest concentration at which the subject identified the taste.
Time Frame: Change from Baseline in threshold of perception at 6 weeks
Measure: Median (Full Range); unit: μmol/ml
Arm/Group | Pre-chemotherapy Patientes | Post-chemotherapy Patients
Number analyzed (Participants) | 40 | 39
μmol/ml | 15.5 [3.5 to 18.5] | 12.5 [3.5 to 18.5]
Statistical Analysis 1: Comparison: Pre-chemotherapy Patientes vs Post-chemotherapy Patients; For the paired analysis of taste acuity we used Wilcoxon for difference between baseline and 6 weeks later; Test type: Superiority or Other; p = 0.608, Wilcoxon (Mann-Whitney)

14. Primary Outcome: Dysgeusia (BITTER Perception)
Description: Describe the perception threshold (PT) of bitter taste with 5 dilutions with different concentrations.
  The patients were instructed to taste each 5 ml dilution in ascending order and to rinse the dilution around the entire oral cavity. After each rinse, the patients were asked whether the sample they took tasted different from water to identify their PT, which was assigned to the lowest concentration at which the subject perceived a difference in taste from water. If so, then the patients were asked to identify the taste to define their RT, which was assigned to the lowest concentration at which the subject identified the taste.
Time Frame: Change from Baseline in threshold of perception at 6 weeks
Measure: Mean (Full Range); unit: μmol/ml
Arm/Group | Pre-chemotherapy Patientes | Post-chemotherapy Patients
Number analyzed (Participants) | 40 | 39
μmol/ml | 97 [91 to 121] | 91 [91 to 121]
Statistical Analysis 1: Comparison: Pre-chemotherapy Patientes vs Post-chemotherapy Patients; For the paired analysis of taste acuity we used Wilcoxon for difference between baseline and 6 weeks later; Test type: Superiority or Other; p = 0.035, Wilcoxon (Mann-Whitney)

15. Primary Outcome: Dysgeusia (BITTER Recognition)
Description: Describe the recognition threshold (RT) of bitter taste with 5 dilutions with different concentrations.
  The patients were instructed to taste each 5 ml dilution in ascending order and to rinse the dilution around the entire oral cavity. After each rinse, the patients were asked whether the sample they took tasted different from water to identify their PT, which was assigned to the lowest concentration at which the subject perceived a difference in taste from water. If so, then the patients were asked to identify the taste to define their RT, which was assigned to the lowest concentration at which the subject identified the taste.
Time Frame: Change from Baseline in threshold of perception at 6 weeks
Measure: Median (Full Range); unit: μmol/ml
Arm/Group | Pre-chemotherapy Patientes | Post-chemotherapy Patients
Number analyzed (Participants) | 40 | 39
μmol/ml | 115 [91 to 121] | 109 [91 to 121]
Statistical Analysis 1: Comparison: Pre-chemotherapy Patientes vs Post-chemotherapy Patients; For the paired analysis of taste acuity we used Wilcoxon for difference between baseline and 6 weeks later; Test type: Superiority or Other; p = 0.402, Wilcoxon (Mann-Whitney)

16. Primary Outcome: Dysgeusia (UMAMI Dilutions Dichotomized)
Description: We divide dilutions in two groups and dichotomized the patients into high and low sensibility to umami taste. (perception)
Time Frame: pre - post chemotherapy (6 weeks)
Measure: Number; unit: participants
Arm/Group | Pre-chemotherapy Patientes | Post-chemotherapy Patients
Number analyzed (Participants) | 40 | 39
participants
  UMAMI 0.3 - 1.5 μmol/ml | 31 | 36
  UMAMI > 1.5 μmol/ml | 9 | 3
Statistical Analysis 1: Comparison: Pre-chemotherapy Patientes vs Post-chemotherapy Patients; for the paired analysis of taste acuity, we used Mc Nemar test for dividing into high and low sensibility to umami, bitter and sweet tastes; Test type: Superiority or Other; p = 0.109, McNemar

17. Primary Outcome: Dysgeusia (SWEET Dilutions Dichotomized)
Description: We divide dilutions in two groups and dichotomized the patients into high and low sensibility to sweet taste.
Time Frame: pre - post chemotherapy (6 weeks)
Population: we dichotomized the patients into high or low sensibility to umami, bitter and sweet tastes pre-postchemotherapy
Measure: Number; unit: participants
Groups:
- Pre-chemotherapy Patientes: patients with high or low sensibility to umami, bitter and sweet tastes pre-chemotherapy
- Post-chemotherapy Patients: patients with high or low sensibility to umami, bitter and sweet tastes post-chemotherapy
Arm/Group | Pre-chemotherapy Patientes | Post-chemotherapy Patients
Number analyzed (Participants) | 40 | 39
participants
  SWEET 3.5 - 9.5 μmol/ml | 26 | 33
  SWEET > 9.5 μmol/ml | 14 | 6
Statistical Analysis 1: Comparison: Pre-chemotherapy Patientes vs Post-chemotherapy Patients; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.092, McNemar

18. Primary Outcome: Dysgeusia (BITTER Dilutions Dichotomized)
Description: We divide dilutions in two groups and dichotomized the patients into high and low sensibility to umami, bitter and sweet tastes
Time Frame: pre - post chemotherapy (6 weeks)
Measure: Number; unit: participants
Arm/Group | Pre-chemotherapy Patientes | Post-chemotherapy Patients
Number analyzed (Participants) | 40 | 39
participants
  BITTER 91 - 103 μmol/ml | 26 | 35
  BITTER > 109 μmol/ml | 14 | 4
Statistical Analysis 1: Comparison: Pre-chemotherapy Patientes vs Post-chemotherapy Patients; We divide dilutions in two groups and dichotomized the patients into high and low sensibility to bitter taste. (PERCEPTION); Test type: Superiority or Other; p = 0.022, McNemar

ADVERSE EVENTS:
Description: Serious and/or Other [non-serious] adverse events were not collected/assessed for this observational study
Groups:
- LUNG CANCER PATIENTS: any toxicity resulting from exposure to chemotherapy with which patients are treated are unrelated to this study, which was observational
Arm/Group | LUNG CANCER PATIENTS
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
No analysis of serum zinc was performed and a small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes